CLINICAL TRIAL: NCT03771430
Title: A Multidisciplinary Intervention in Total Knee Arthroplasty - a Multicenter, Randomized Controlled Trial in OA Patients (The MultiKnee Trial)
Brief Title: A Multidisciplinary Intervention in Total Knee Arthroplasty
Acronym: MultiKnee
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lovisenberg Diakonale Hospital (Other)
Collaborators: Haukeland University Hospital (Other); Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MultiKnee Trial
Record Dates: First submitted 2018-11-12; First posted 2018-12-11 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-06

CONDITIONS: Osteoarthritis; Primary; Degenerative Joint Disease of Knee
Keywords: Total knee arthroplasty; Physiotherapy; Cognitive behavioral therapy; e-therapy
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee | interventions — Exercise; Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-surgical group (Experimental): Osteoarthritis education, exercise and eCBT
  Interventions: Behavioral: Osteoarthritis education, exercise and CBT
- Combined group (Experimental): Total knee arthroplasty + osteoarthritis education, exercise and eCBT
  Interventions: Behavioral: Osteoarthritis education, exercise and CBT; Procedure: Total Knee Arthroplasty
- Surgery only (standard care) (Active Comparator): Total knee arthroplasty + standard physiotherapy
  Interventions: Procedure: Total Knee Arthroplasty

INTERVENTIONS:
Behavioral: Osteoarthritis education, exercise and CBT — Osteoarthritis Education
  1. 60-min session by AktivA trained PT)
     * Signs/symptoms, risk factors, weight control, treatment
     * Importance of physical activity
     * Appropriate activity & training modalities
     Exercise and CBT Support
  2. 60-min sessions/week for 12 weeks (a total of 24 sessions) led by AktivA and CBT trained PT)
     * Warm-up session
     * Strengthening exercises
     * Functional exercises
     * Stretching
     * Monitoring of CBT progress
     * Review of CBT lessons learned
     * Integration of CBT skills
     * Enhance motivation to continue
  Online CBT (iCBT) (10 modules completed at home)
  * Pain causes & prevention
  * Pain management
  * Health promotion & stress reduction at home & work
  * Adapting for leisure & work
  * Controlling flare-ups
  * Maintaining & improving results
  Other Names: AktivA
  Arms: Combined group; Non-surgical group
Procedure: Total Knee Arthroplasty — Standard total knee arthroplasty will be performed.
  Other Names: knee replacement
  Arms: Combined group; Surgery only (standard care)

SUMMARY:
The purpose of this study is to investigate the effectiveness of cognitive behavioral therapy delivered as an e-therapy program, combined with physical exercise delivered by physiotherapists, for patients on waiting list for total knee arthroplasty. The patients will be randomized to either 1) a non-surgical program consisting of web-based cognitive behavioral therapy combined with physiotherapy, 2) total knee arthroplasty (TKA) surgery followed by web-based cognitive behavioral therapy combined with physiotherapy, or 3) a control group who undergo TKA followed by standard physiotherapy.

DETAILED DESCRIPTION:
The study is a multidisciplinary trial testing an intervention delivered by physiotherapists. Up to 20% of total knee arthroplasty (TKA) patients continue to experience moderate/severe pain 12 months after TKA. While physical therapy (PT) and cognitive-behavior therapy (CBT) have shown promise for improving outcomes, they have not been evaluated in combination or in patients at risk for chronic pain after TKA. This trial will evaluate PT+CBT combined, either as a substitute for or as a supplement to TKA for patients at risk for chronic pain after TKA.

Pilot/Feasibility study:

The study will include a feasibility/pilot study with 15 patients to be performed from November 2018. The intervention and study procedures may be modified based on results from the feasibility/pilot study.

Full scale Randomized Controlled Trial (RCT):

The full-scale RCT will include 282 patients scheduled for TKA. Patients will be randomly assigned to one of three groups: 1) non-surgical intervention (i.e., PT+CBT), 2) a combination of TKA with pre- and postoperative PT+CBT, or 3) A control group receiving TKA and usual care follow-up. Primary outcome: The Pain subscale from the KOOS. The intervention has the potential to improve outcomes for patients who currently obtain little benefit from standard TKA.

Cross-sectional observational study: Patients declining to participate in the RCT will be offered the option to participate in a separate cross-sectional study. The inclusion and exclusion criteria will be identical to the RCT. Patients who agree to participate in the cross-sectional study will complete the same baseline questionnaires as in the RCT and are asked about the reasons they did not want to participate in the RCT.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for TKA for OA at Lovisenberg, Oslo; Martina Hansen, Bærum, or Coastal Hospital Hagevik, Bergen
2. Age 18 - 79 years
3. ASA grade 1-3
4. KL grade 3 or 4
5. BMI<40
6. Able to read and write in Norwegian

Exclusion Criteria:

* Diagnosis of dementia or sero-positive rheumatic disease
* Previously undergone uni or patellofemoral prosthesis in the index knee
* Large axis deviation or instability requiring use of hinged implants
* Scheduled for unicompartmental arthroplasty or revision surgery

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2019-08-28 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in the knee injury and osteoarthritis score (KOOS) pain subscale | Before randomization, 12 months after treatment start. Also measured at 3, 6, and 24 months after treatment start.12 months after treatment start will be the primary outcome.
  KOOS is a knee-specific, patient administered questionnaire developed to evaluate short- and long-term symptoms and functioning in subjects with knee injury and osteoarthritis. KOOS is validated for use in total knee arthroplasty and has been shown to be a valid, reliable and responsive measure. KOOS is a patient-administered questionnaire.
  The KOOS is a knee joint specific questionnaire with 42 items designed to assess patients' opinions about their difficulties with activity due to problems with their knees during the past week. The pain subscale of the KOOS consists of 9 items that assess frequency of pain and pain severity in different situations. Each of the 42 items carries equal weighting (0-4), with higher scores indicating better functioning. The pain subscale score will be transformed to a 0-100 scale, with 0 representing extreme knee problems and 100 representing no problems.

SECONDARY OUTCOMES:
Knee injury and osteoarthritis score (KOOS) subscores: Other symptoms, activities of daily living (ADL), function in sport and recreation, and knee-related quality of life (QOL) | Before randomization. 3, 6, 12 and 24 months following treatment start
  KOOS is a knee-specific questionnaire developed to evaluate short- and long-term symptoms and functioning in subjects with knee injury and osteoarthritis.
  The KOOS is a knee joint specific questionnaire with 42 items designed to assess patients' opinions about their difficulties with activity due to problems with their knees during the past week. KOOS has 5 subscales: pain, other symptoms, activities of daily living (ADL), function in sport and recreation, and knee-related QOL. The KOOS has been validated for use in TKA and has been shown to be valid, reliable and responsive. Each of the 42 items carries equal weighting (0-4), with higher scores indicating better functioning. Each of the subscale scores are transformed to a 0-100 scale, with 0 representing extreme knee problems and 100 representing no problems. KOOS is a patient-administered questionnaire.
The 30 second sit to stand test | Before treatment start. 3, 6, 12 and 24 months following treatment start
  The 30-second sit to stand test will be used to assess functional lower extremity strength. This test is performed using a chair of standard height without arms. The participant is encouraged to complete as many full stands as possible within 30 seconds.
Brief Pain inventory | Before randomization. 3, 6, 12 and 24 months following treatment start
  The Brief Pain Inventory (BPI) will be used to measure pain (56). The BPI is a brief patient-completed questionnaire that consists of four items that measure pain intensity (on an 11-point numeric rating scale from 0-10), seven questions on pain interference with functioning, a body map to localize the pain and one item on pain relief.
EuroQol-5D-5L | Before randomization. 3, 6, 12 and 24 months following treatment start
  The widely used EuroQol-5 (EQ-5D-5L) will be used to measure health-related quality of life.
  The EQ5D-5L consists of two parts: A descriptive system (Mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and the EQ-VAS that record patients self-rated health on a visual analog scale that range from 0 - 100, higher levels indicate better self-rated health.
  The descriptive system can be converted to a single summary index number where lower levels indicate poorer health-related quality of life.
The Forgotten Joint Score | Before randomization. 3, 6, 12 and 24 months following treatment start
  The Forgotten Joint Score will be used to assess how natural the prosthesis feels after total knee arthroplasty. The scoring system consists of 12 items that assess patients agreement with 12 statements, that range from 1 (never) to 5 (mostly). The raw score is transformed to a 0-100 score and then reversed to obtain the final score. A higher score indicate better outcome.
Pain Catastrophizing Scale | Before randomization. 3, 6, 12 and 24 months following treatment start
  The Pain Catastrophizing scale (PCS) will be used to measure catastrophic thinking related to pain. The scale consist of 13 items that range from 0 -4. The PCS assesses three dimensions of catastrophizing (i.e., rumination (range 0-16), magnification (range: 0-12, helplessness (range 0 -24). Higher scores indicate higher levels of catastrophic thinking related to pain. A total score can be computed by summing responses to all 13 items. PCS total scores range from 0-52. Higher scores indicate higher levels of catastrophic thinking related to pain.
Patient-acceptable symptom state, perceived treatment failure. | At 3, 6, 12 and 24 months following treatment start.
  Patient-acceptable symptom state will be measured by a single item question. The patient state wether they consider their knee function satisfactory or not (Yes/No).
  Perceived treatment failure will be measured by a single item question. The patient state whether their situation is so dissatisfying that they consider the treatment as a failure (Yes/No).
Global perceived effect | At 3, 6, 12 and 24 months following treatment start.
  The patient rate their level of knee problems compared to their condition before they started their treatment, by choosing on of seven statements that describe the level of improvement/worsening.
  The statements range from "better - an important improvement" - to "worse, an important worsening".
Adverse events/serious adverse events | From treatment start until 24 months following treatment start.
  All events reported by participant, physiotherapist or documented in the patient's hospital record.
  * During surgery: Number of patients with fractures (Tibia, patella, femur), nerve or vascular injury, rupture of patella tendon, other.
  * Postoperatively: Number of patients with deep infection, any secondary surgery (e.g., skin necrosis or scar tissue adherences, DAIR, MUA, secondary insertion of patella component, partial/total revision surgery), supracondylar femur fracture, patella fracture, permanent n. peroneus paresis, aseptic loosening, polyethylene defect (tibia or patella), instability requiring intervention, thrombophlebitis demanding anticoagulant treatment, pulmonary embolism, myocardial infarction, cerebral insult, other events.
  * Patient-reported myocardial infarction, cerebral insult, pulmonary embolism or DVT within 3 months following intervention.
  * All events reported by patients or physiotherapists - open probe questionnairing

OTHER OUTCOMES:
Pittsburgh Sleep Quality Index | Before randomization. 3, 6, 12 and 24 months following treatment start
  The Pittsburgh Sleep Quality index (PSQI) is a widely-used self-report measure of sleep disturbance during the past month. The PSQI consists of 19 items that measures different aspects of sleep. The 19 items produce 7 component scores (i.e., duration of sleep, sleep disturbance, sleep latency, day dysfunction due to sleepiness, sleep efficiency, overall sleep quality, need for sleep medications) each ranging from 0-3 where higher score indicate poorer sleep. All component scores can be summarized to a global score that range from 0 to 21 where higher scores indicate poorer sleep quality. The PSQI has good validity and reliability.
The Hospital Anxiety and Depression Scale | Before randomization. 3, 6, 12 and 24 months following treatment start
  The Hospital Anxiety and Depression Scale (HADS) will be used to measure self-reported psychological distress (depression and anxiety). The scale consists of 14 items, 7 on the depression subscale and 7 on the anxiety subscale. The Norwegian version has excellent psychometric properties. Each subscale range from 0-21 where higher scores indicate higher levels of anxiety or depression. A total score (range 0 - 42) can be calculated from summarizing all the 14 items. Higher scores indicate higher levels of anxiety/depression.
The Fear-Avoidance Belief Questionnaire | Before randomization. 3, 6, 12 and 24 months following treatment start
  The Fear-Avoidance Belief Questionnaire (FABQ) will be used to measure pain-related fear of movement. The instrument consists of 2 subscales, fear-avoidance beliefs for work, and fear-avoidance beliefs for physical activity (FABQ-PA). Only the FABQ-PA subscale will be used in this study. The FABQ-PA consists of 4 items where patients rate their agreement with 5 statements about pain and physical activity. The FABQ-PA range from 0-24 and higher scores indicate higher levels of pain-related fear of movement.
Health Locus of Control Scale | Before randomization. 3, 12 and 24 months following treatment start
  The Health Locus of Control Scale (HLCS) will be used to measure patients' anticipations between own health and disease behavior and consequences of the behavior. The scale consists of 18 statements. Patients rate their agreement on a 6 point likert scale ranging from disagrees completely to agrees completely. Scoring: The scoring system consists of 3 subscales: The Internal Locus of Control, the Powerful Others Health Locus of Control, and the Chance Health Locus of control. The scores are obtained by summing items for each subscale. Higher scores indicate stronger agreement or inclination towards that particular subscale.
Self-reported level of physical activity | Before randomization. 3, 6, 12 and 24 months following treatment start
  Self-reported level of physical activity will be measured using two items from the Norwegian Hunt2 survey that assess frequency of light and hard physical activity, and the Stages of Change for physical activity. The Stages of Change for physical activity assess patients' readiness for physical activity. Patients rate their agreement with five different statements about physical activity.
The ActiGraph Professional single-axis accelerometer | Before treatment start. 6, 12 and 24 months following treatment start
  The ActiGraph Professional single-axis accelerometer, a body worn sensor system to measure physical activity, will be used to measure time in sedentary and active positions, duration of activity and number of steps during walking
The 40 meters walk test | Before treatment start. 3, 6, 12 and 24 months following treatment start
  The 40 meter walk test: The patient is instructed to walk 40 meter under timing.
Stair Climb Test | Before treatment start. 3, 6, 12 and 24 months following treatment start
  The Stair Climb Test will be used to measure ascending and descending stair activity, and lower body strength and balance, measured as a participants' time in seconds to ascend and descend a flight of stairs.
Registry-based data on use of health care resources | From before randomization until 3, 6, 12 and 24 months after treatment start.
  Use of health care resources will be measured using registry data from the KUHR-system (i.e., control and payment of reimbursements to health service providers), the Norwegian Patient Registry (NPR) FD Trygd social security database, the Norwegian Prescription Database and the Norwegian Arthroplasty registry. All information will be anonymized and linked to each patient using a code number before analysis.
Radiographs: weightbearing AP, lateral view, Rosenberg view and long leg weightbearing AP view (HKA) | Before treatment start, 12 months following treatment start.
  X-rays including weightbearing AP, lateral view, Rosenberg view and long leg weightbearing AP view (HKA) weightbearing AP view (HKA). OA severity grading will be performed according to the Kellgren-Lawrence grading system and cartilage thickness.
Screening and recruitment of patients (pilot study with 15 patients). | Baseline T1 before randomization
  Number of patients undergoing screening, considered for inclusion, eligible for inclusion, consenting to participate and undergoing randomization
Adherence to the intervention (pilot study with 15 patients) | From treatment start until 12 weeks following treatment start.
  Number of patients receiving the full dose of the intervention. adverse events, recruitment, screening and randomization, retention in study/loss to follow-up.
Acceptability of the intervention (pilot study with 15 patients) | From treatment start until 12 weeks following treatment start.
  Number of patients feeling overwhelmed or burdened by the intervention. Number of patients not completing the intervention due to feeling overwhelmed ro burdened by the intervention.
Level of electronic health literacy | Before treatment start, 6 months after treatment start
  The Electronic Health Literacy Questionnaire (e-HLQ) (44) will be used to measure patients level of electronic health literacy prior to, and six months following surgery. In this study, 4 domains will be assessed: 1) using technology to process health information, 2) understanding of health concepts and language, 3) ability to actively engage with digital services, 4) motivated to engage with digital services. The scores range 1-4, with high scores indicating high e-health literacy.
Level of health literacy | Before treatment start, 6 months after treatment start
  The International Health Literacy Population survey Questionnaire 2019-2021(HLS19-Q47) will be used to measure patients' level of health literacy prior to, and six months following surgery. The original HLS-19-Q47 consist of 47 items. In this study, 2 domains will be assessed: 1) Health promotion and 2) General health literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Anners Lerdal, PhD, Principal Investigator — Lovisenberg Diaconal Hospital, University of Oslo; Arild Aamodt, PhD, Principal Investigator — Lovisenberg Diakonale Hospital; Maren F Lindberg, PhD, Study Director — Lovisenberg Diakonale Hospital/University of Oslo; Kari Indrekvam, PhD, Study Chair — Haukeland University Hospital - Kysthospitalet Hagevik/University of Bergen; Stig Heir, PhD, Study Chair — Martina Hansens Hospital
Locations (3):
- Norway (3):
  - Haukeland University Hospital - Kysthospitalet Hagevik, Bergen
  - Lovisenberg Diaconal Hospital, Oslo
  - Martina Hansens Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kise NJ, Eliassen S, Furnes O, Gay C, Heir S, Lerdal A, Lindberg MF, Rognsvag T, Aamodt A, Nerhus TK. Fear avoidance and catastrophizing are associated with both knee awareness and quality of life in knee osteoarthritis patients: a secondary report of a cross-sectional study. Acta Orthop. 2025 Dec 18;96:920-926. doi: 10.2340/17453674.2025.45070. PMID 41410384
- [Derived] Rognsvag T, Bergvad IB, Furnes O, Indrekvam K, Lerdal A, Lindberg MF, Skou ST, Stubberud J, Badawy M. Exercise therapy, education, and cognitive behavioral therapy alone, or in combination with total knee arthroplasty, in patients with knee osteoarthritis: a randomized feasibility study. Pilot Feasibility Stud. 2024 Feb 28;10(1):43. doi: 10.1186/s40814-024-01470-y. PMID 38419024
- [Derived] Lindberg MF, Aamodt A, Badawy M, Bergvad IB, Borchgrevink P, Furnes O, Gay C, Heir S, Holm I, Indrekvam K, Kise N, Lau B, Magnussen J, Nerhus TK, Rognsvag T, Rudsengen DE, Rustoen T, Skou ST, Stubberud J, Smastuen MS, Lerdal A. The effectiveness of exercise therapy and education plus cognitive behavioral therapy, alone or in combination with total knee arthroplasty in patients with knee osteoarthritis - study protocol for the MultiKnee trial. BMC Musculoskelet Disord. 2021 Dec 20;22(1):1054. doi: 10.1186/s12891-021-04924-z. PMID 34930194
- [Derived] Rognsvag T, Lindberg MF, Lerdal A, Stubberud J, Furnes O, Holm I, Indrekvam K, Lau B, Rudsengen D, Skou ST, Badawy M. Development of an internet-delivered cognitive behavioral therapy program for use in combination with exercise therapy and education by patients at increased risk of chronic pain following total knee arthroplasty. BMC Health Serv Res. 2021 Oct 25;21(1):1151. doi: 10.1186/s12913-021-07177-7. PMID 34696785